CLINICAL TRIAL: NCT02024048
Title: Evaluation of Choroidal Thickness During Pregnancy Using Enhanced Depth Imaging Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gaia Hospital (Other)
Responsible Party: Principal Investigator, Renata Rothwell, Dr, Gaia Hospital
Other Study IDs: ECTP-EDI
Record Dates: First submitted 2013-12-18; First posted 2013-12-31 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Pregnancy
Keywords: Pregnancy; OCT; Enhanced depth imaging; Choroid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregnant: OCT
  Interventions: Other: OCT
- Control: OCT
  Interventions: Other: OCT

INTERVENTIONS:
Other: OCT — Optical coherence tomography in enhanced depth imaging mode

SUMMARY:
The purpose of this study is to evaluate choroidal thickness and volume during the third trimester of pregnancy by comparison with a group of age-matched non-pregnant healthy group of women

DETAILED DESCRIPTION:
Pregnant women in the last trimester and age-matched healthy controls have an Optical Coherence Tomography (OCT) image taken on the OCT Spectralis® device.

A map of the choroid in the macular area is constructed automatically. Choroidal thickness and volume are calculated for the 9 subfields defined by the Early Treatment Diabetic Retinopathy Study (ETDRS).

A comparative analysis between the two groups will be performed. As a secondary outcome measure, the change in choroidal thickness of the pregnant group of women will be assessed at 6 months postpartum by comparison to the 3rd trimester of pregnancy.

The OCT is a non-invasive examination that poses no risk to the mother or the fetus.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women:

* uncomplicated pregnancy in the third trimester (from 28 weeks of gestation)

For both groups:

* no systemic or ocular disease
* absence of systemic medication other than prenatal vitamins
* no smoking habits
* emmetropia or a small refractive error (spherical equivalent <1.5 diopters)

Exclusion Criteria:

* any of the above

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy pregnant women in the third trimester of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Choroidal thickness | 3rd trimester of pregnancy (from 28 weeks gestation to delivery)
  Comparison of choroidal thickness between the pregnant group of women and the age-matched group of control subjects

SECONDARY OUTCOMES:
Change in choroidal thickness | During the 3rd trimester (from 28 weeks gestation to delivery) and at 6 months post partum
  Change in choroidal thickness in the third trimester of pregnancy and at 6 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Renata Rothwell, Dr, Principal Investigator — Department of Opthalmolgy, Centro Hospitalar Vila Nova de Gaia/Espinho; Sofia Fonseca, Dr, Principal Investigator — Department of Ophthalmology, Centro Hospitalar Vila Nova de Gaia/Espinho; Marisa Oliveira, Dr, Principal Investigator — Department of Ophthalmology, Centro Hospitalar Vila Nova de Gaia/Espinho; Lígia Ribeiro, Dr, Principal Investigator — Department of Ophthalmology, Centro Hospitalar Vila Nova de Gaia/Espinho; Dália Meira, Dr, Principal Investigator — Department of Ophthalmology, Centro Hospitalar Vila Nova de Gaia/Espinho
Locations (1):
- Department of Ophthalmology, Centro Hospitalar Vila Nova de Gaia/Espinho Vila Nova de Gaia, Vila Nova de Gaia, Portugal